CLINICAL TRIAL: NCT02469974
Title: Ruxolitinib in Combination With High Dose Therapy and Autologous Stem Cell Transplantation for Myelofibrosis
Brief Title: Ruxolitinib in Combination With Autotransplant
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no enrollments
Sponsor: Marina Kremyanskaya (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor-Investigator, Marina Kremyanskaya, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 14-2106
Record Dates: First submitted 2015-05-28; First posted 2015-06-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Myelofibrosis; MF
Keywords: Myelofibrosis; RUXOLITINIB; Autologous stem cell transplant
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib; Filgrastim; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ruxolitinib / INC 424 (Experimental): Ruxolitinib, Jakafi ®, will be given orally at standard dose daily for 16 weeks pre ASCT and up to 3 months post-ASCT for 10 patients (allowing for 2 additional screen failures). Patients will restart ruxolitinib at 100 days after the ASCT as long as their platelet count is at least 50 x103. For patients whose platelet count is below 50 x103 at day 100, ruxolitinib should be restarted once platelet count reaches 50 x103. The dose of ruxolitinib can be titrated up as per clinical guidelines. PBSC mobilization will include G-CSF 10 mcg/kg/day. HDC for ASCT will consist of IV busulfan 2.0 mg/KBW once daily x 4 for days -5 to -2.
  Interventions: Drug: RUXOLITINIB / INC 424; Drug: Filgrastim; Drug: Busulfan

INTERVENTIONS:
Drug: RUXOLITINIB / INC 424 — Administered orally 5-20 mg twice daily x 16 weeks of therapy prior to attempted peripheral blood stem cells (PBSC) collection, during the collection and rest period and 3 months of therapy after high dose chemotherapy (HDC).
  Other Names: RUX; Jakafi®
Drug: Filgrastim — Peripheral blood stem cells (PBSC) will be mobilized with filgrastim 10 mcg/kg/day IV
  Other Names: Neupogen®
Drug: Busulfan — Conditioning for autologous Hematopoeitic Stem Cell Transplantation (HSCT) will consist of IV busulfan 2.0 mg/KBW once daily x 4 for days -5 to -2
  Other Names: Busulfex®

SUMMARY:
To determine the safety of the approach of giving RUXOLITINIB before and after an autologous stem cell transplant, as measured by graft failure or death.

DETAILED DESCRIPTION:
This is a pilot, single arm, single center study with no stratification to assess the safety (measured by graft failure or death) and feasibility (measured by adequacy of stem cell collection) of combining ruxolitinib with autologous Hematopoeitic Stem Cell Transplantation (HSCT) in patients with advanced myelofibrosis (MF). Patients will receive a short course of ruxolitinib prior to and during mobilization of HSCT with Filgrastim. Conditioning for the autologous HSCT will consist of Bulsulfan. Post-transplant patients will receive ruxolitinib maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented diagnosis of MF (idiopathic or post PV/ET)
* Age 18-75 years
* Intermediate-2/ high-risk disease as per Dynamic IPSS (DIPSS) criteria or Intermediate-1 risk disease with one of the following features within one year from screening:

  1. Red cell transfusion dependency
  2. unfavorable Karyotype
  3. platelet count <100 x 109/L
  4. symptomatic splenomegaly
  5. PB blasts > 1%
  6. Blasts in PB <20% prior to study enrollment
  7. No available suitable matched related (6/6 or 5/6) or unrelated donor (8/8 or 7/8 allele matched) or unwilling or unable to pursue allogeneic stem cell transplant
  8. WBC <50,000/ml at screening
* Able to give informed written consent
* ECOG Performance status of 0-2
* Life expectancy >6 months
* Off all myelofibrosis-related investigational or standard agents (except for ruxolitinib) for at least 4 weeks prior to study enrollment and recovered from all toxicities. If patient is already on ruxolitinib for a minimum of 16 weeks prior to study enrollment, patient can proceed to mobilization and collection
* Adequate organ function defined as the following (*unless clearly disease related):

  1. Adequate renal function - creatinine <2 x ULN
  2. Adequate hepatic function - AST/ALT <3 x ULN, Total Bilirubin <3 x ULN, exception is elevated indirect bilirubin attributed to Gilbert's syndrome or hemolysis
  3. Adequate hematopoietic function - Platelet ≥50 x 109/L (without transfusion) and ANC ≥1.0 x 109/L
  4. LVEF >40% (MUGA or echocardiogram)
  5. Adequate pulmonary function with DLCO >40%

Exclusion Criteria:

* Hypersensitivity to JAK inhibitor
* Clinical evidence of cirrhosis
* Leukemic transformation (>20% blasts in PB or BM any time prior to HCT)
* Platelet count <50 x 109/L
* Active uncontrolled infection
* History of another malignancy within 5-years of date of HCT except history of basal cell or squamous cell carcinoma of skin or PV or ET
* Known HIV positive
* Woman of childbearing potential unwilling or unable to use adequate contraception Pregnant or nursing females Known active infection with hepatitis A, B or C virus

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Safety of combining ruxolitinib with autologous HSCT measured by graft failure or death | 2 years
  Safety of this approach as measured by graft failure or death

SECONDARY OUTCOMES:
CD34 cells | 4 years
  Total CD34+ cell dose will be calculated based on results of flow cytometric analysis and patient's weight.
The regimen related mortality (RRM) | day 100
The regimen related mortality (RRM) | day 365
Rate of engraftment/graft failure | 4 years
Time of engraftment for neutrophils and platelets | 4 years
The incidence of serious infectious complications | up to 1 year post transplant
Changes in marrow fibrosis score | at 180 and 365 days post-transplant
  The myelofibrosis score will be assessed as per the European Consensus Grading published by Thiele Grading Description at 365 days as compared to 180 days
Change in FISH allele | at 365 days post-transplant
  Changes in FISH abnormalities when present will be measured by cytogenetics.
Change in JAK allele | at 365 days post-transplant
  Changes in Jak 2 V617F allele burden when present will be measured by quantitative RT-PCR
Rate of response | at 6 months post-transplant
  Overall efficacy will be rated on a scale as complete remission, partial remission, clinical improvement, or stable disease
Rate of response | at 1 year post-transplant
  Overall efficacy will be rated on a scale as complete remission, partial remission, clinical improvement, or stable disease

CONTACTS AND LOCATIONS:
Overall Officials: Marina Kremyanskaya, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai